CLINICAL TRIAL: NCT05201976
Title: A Clinical Trial Investigating the Effects of a Virtually Implemented Home Based Cardiac Rehab Program with Real-time, Video-based Exercise Supervision and Vitals Monitoring
Brief Title: Effect of a Virtually Implemented Cardiac Rehabilitation Program
Acronym: VIRT-CR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Independence Blue Cross (Other); CardaHealth (Unknown)
Responsible Party: Principal Investigator, Neel Chokshi, Principal Investigator, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 848902
Record Dates: First submitted 2021-12-05; First posted 2022-01-21 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Randomized, non-inferiority, Case vs. Control (1 to 1)
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Active Comparator): Virtual cardiac rehab program delivered through the CardaHealth platform.
  Interventions: Other: Virtually administered Cardiac Rehab program
- Control (Active Comparator): Clinically ordered standard of care cardiac rehab program (in-person).
  Interventions: Other: Standard of Care in person Cardiac Rehab Program

INTERVENTIONS:
Other: Virtually administered Cardiac Rehab program — Virtual cardiac rehab program delivered through the CardaHealth platform.
  Arms: Intervention
Other: Standard of Care in person Cardiac Rehab Program — Clinically ordered standard of care cardiac rehab program (in-person).
  Arms: Control

SUMMARY:
A clinical trial investigating the effects of a virtually implemented home-based cardiac rehab program with real-time, video based exercise supervision and vitals monitoring.

DETAILED DESCRIPTION:
This study will use a randomized, controlled trial design to test the effectiveness of a virtually implemented cardiac rehabilitation (CR) program with real-time, video based supervised exercise and vitals monitoring as compared to traditional center based rehab in patients with a clinical indication for cardiac rehab. The primary outcome of effectiveness will be change in cardiorespiratory fitness as assessed by maximal VO2 achieved at the start of CR and on upon completion of CR.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been prescribed cardiac rehabilitation as part of their standard of care

Exclusion Criteria:

* Patients with significant exercise limitations other than cardiovascular disease
* Patients who are unable to exercise in home
* Patients with active cancer treatment
* Patients who do not have an email address or a cell phone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2021-11-08 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2024-10-15 (Actual)

PRIMARY OUTCOMES:
Change in VO2 max (ml/kg/min) | At baseline visit and at the end of study approximately 40 weeks
  Cardiorespiratory fitness as assessed by maximal VO2

SECONDARY OUTCOMES:
Attendance | Mean number of cardiac rehab sessions completed per patient, over the course of 12 weeks or 36 sessions.
  Subject's adherence to scheduled cardiac rehab sessions.
Quality of Life questionnaire | Prior to beginning of cardiac rehabilitation and then at completion of cardiac rehabilitation program approximately 36 weeks
  Subject's completion of SF-36
Blood Pressure | Start of each cardiac rehab session, over the course of 12 weeks or 36 sessions.
  Change in systolic and diastolic blood pressure over the duration of the study. BP will be self-assessed by the subjects at the start of each session.
Major adverse cardiovascular events (MACE) | Events will be collected up to 27 months post study enrollment
  Major cardiovascular events include cardiovascular hospitalizations and mortality
Survey | At completion of cardiac rehabilitation program approximately 36 weeks
  Patient satisfaction, physician satisfaction
Change in LDL | Labs will be collected up to 27 months post study enrollment
  Ascertained through the electronic health through routinely collected values
Change in HDL | Labs will be collected up to 27 months post study enrollment
  Ascertained through the electronic health through routinely collected values
Change in triglycerides | Labs will be collected up to 27 months post study enrollment
  Ascertained through the electronic health through routinely collected values

CONTACTS AND LOCATIONS:
Overall Officials: Srinath Adusumalli, MD, Principal Investigator — University of Pennsylvania; Neel Chokshi, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No